CLINICAL TRIAL: NCT05599542
Title: The Effect of Hypno-breastfeeding and Solution-oriented Approach on Mothers' Breastfeeding Motivation and Perception of Insufficient Milk: Randomize Controlled Study
Brief Title: The Effect of Hypno-breastfeeding and Solution-oriented Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Elif DAĞLI, Lecturer Doctor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: hypno-breastfeeding
Record Dates: First submitted 2022-10-03; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Breastfeeding; Breast Milk Expression
Keywords: Hypno-breastfeeding; Solution-oriented approach
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Solution-oriented approach group (Experimental): A preliminary assessment of the pregnant woman's thoughts on breastfeeding was made and the EARS (Eliciting, Amplifying, Reinforcing and Start Over) process was applied. Eliciting, Amplifying, Reinforcing and Start Over process guides the second and subsequent sessions in a sequential order.
  Interventions: Other: Solution-oriented approach; Other: Hypno-breastfeeding
- Hypno-breastfeeding group (Experimental): A preliminary assessment was made about the pregnant woman's thoughts on breastfeeding. In the hypno-nursing philosophy, affirmation, relaxation, imagination and visualization techniques were used in order to positively affect the subconscious mind during the breastfeeding process.
  Interventions: Other: Solution-oriented approach; Other: Hypno-breastfeeding
- control group (Other): Data were collected with the Introductory Information Form at the first interview (admission to the postpartum service) with the women in the control group. Post-test data were collected with Primiparous Breastfeeding Motivation Scale and Insufficient Milk Perception Scale at 16-24 hours postpartum.
  Interventions: Other: Solution-oriented approach; Other: Hypno-breastfeeding

INTERVENTIONS:
Other: Solution-oriented approach — A preliminary assessment of the pregnant woman's thoughts on breastfeeding was made and the EARS (Eliciting, Amplifying, Reinforcing and Start Over) process was applied. Eliciting, Amplifying, Reinforcing and Start Over process guides the second and subsequent sessions in a sequential order. The Eliciting, Amplifying, Reinforcing and Start Over technique reminds the counselor of the basic concepts of solution-oriented approach and its explanation is as follows;
Other: Hypno-breastfeeding — A preliminary assessment was made about the pregnant woman's thoughts on breastfeeding. In the hypno-nursing philosophy, affirmation, relaxation, imagination and visualization techniques were used in order to positively affect the subconscious mind during the breastfeeding process.

SUMMARY:
Motivation, which is also necessary for the breastfeeding behavior of mothers in the postpartum period, can affect the success and continuity of breastfeeding. This study was conducted to evaluate the effects of hypno-breastfeeding and solution-oriented approach on breastfeeding motivation and insufficient milk perception in mothers. It is a randomized controlled experimental study. The sample of the study consisted of 90 women who met the inclusion criteria, three groups as the hypno-breastfeeding group, the solution-focused approach group and the control group.

DETAILED DESCRIPTION:
Hypno-breastfeeding, which is a mind-body program that helps to increase breast milk production, is a therapy that includes emotion control, pain management, and positive suggestions that define the mother's role in the breastfeeding process. This method, in comfortable, calm and natural conditions, is effective in increasing the amount of milk by eliminating phobias, anxiety and negative thoughts in the mind of the mother, relaxing and concentrating on breastfeeding. The solution-oriented approach, on the other hand, is a therapeutic counseling practice that does not deal with the problem itself, but focuses on the past successes of the individual and the times when they did not experience the problem. In solution-oriented approach, which argues that each individual can solve their problems with their own internal resources by only directing them to the positive, it focuses on the strengths of the person instead of underlining the weaknesses. No study has been found on the effect of solution-oriented approach on breastfeeding process in the perinatal period. However, there are studies that show that the application of solution-oriented approach, which will make a different contribution to midwifery philosophies, is effective in reducing the fear of birth and reducing the anxiety of mothers who have anxiety about premature baby care. It is thought that with the effective use of the hypno-breastfeeding method and solution-oriented approach by midwives and health personnel, the perception of insufficient milk of mothers during the breastfeeding process can be reduced and breastfeeding motivation will be positively affected. In this context, this study aimed to determine the effect of hypno-breastfeeding and solution-oriented approach on breastfeeding motivation and insufficient milk perception.

ELIGIBILITY:
Inclusion Criteria:

* Single pregnancy
* 35 weeks and above healthy pregnancy
* No communication barrier
* No diagnosed psychiatric problem
* Normal delivery
* No complications of mother and baby

Exclusion Criteria:

* Multiple pregnancy
* 34 weeks and below pregnancy
* Communication barrier
* Clinical diagnosis of psychiatric problem
* Cesarean delivery
* Complications in mother and baby

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 90 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Primiparous Breastfeeding Motivation Scale | 5 months
  The scale, which was validated and reliable in Turkish by Akçay and Demirgöz Bal, was developed by Stockdale et al. to determine the factors affecting breastfeeding motivation in primiparous women. It was determined that the scale consisting of 29 items was 7-point Likert type and had 4 sub-dimensions. These sub-dimensions are: the value attached to breastfeeding, self-efficacy, perceived midwife support, and success expectancy. As the score obtained from each sub-dimension increases, the breastfeeding motivation level of that sub-dimension increases. A cutoff in the assessment of the scale There is no value or total score. Evaluation by summing the scores obtained in each subgroup in the scale is done. As the score increases, the characteristics of the subgroup and therefore the motivation increase.

SECONDARY OUTCOMES:
Insufficient Milk Perception Scale | 5 months
  The scale, developed by McCarter-Spaulding, consists of 6 questions to determine inadequate perception of breast milk. The Turkish validity and reliability of the scale was performed by Gökçeoğlu. The first question of the scale questions whether the mother perceives her milk adequately and is answered as "yes" or "no". Other questions of the scale are aimed at measuring the perception of inadequacy of milk. These questions are scored between 0-10 ("0" is perceived as completely inadequate, "10" is perceived as completely sufficient). A score between 0-50 can be obtained from the scale, and a high total score indicates an increased perception of milk sufficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Feyza Aktaş Reyhan, Dr., Study Chair — Kütahya Health Sciences University
Locations (1):
- Çukurova University, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No